CLINICAL TRIAL: NCT00793000
Title: A Phase 1 Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-04287881 After First Time Administration Of Ascending Single Oral Doses To Healthy Adult Subjects
Brief Title: Safety And Pharmacokinetics Study Of PF-04287881 In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B0581001
Record Dates: First submitted 2008-11-12; First posted 2008-11-18 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Respiratory Tract Infections
Keywords: Safety tolerability pharmacokinetics PK first in human FIH
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 2 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 3 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 4 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 5 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 6 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 7 (Experimental)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 8 (Experimental): Japanese volunteers, low dose previously tested (based on PK)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 9 (Experimental): Japanese volunteers, intermediate dose previously tested (based on PK)
  Interventions: Drug: PF-04287881; Drug: Placebo
- Cohort 10 (Experimental): Japanese volunteers, high dose previously tested (based on safety)
  Interventions: Drug: PF-04287881; Drug: Placebo

INTERVENTIONS:
Drug: PF-04287881 — 75 mg oral dose (prepared solution) given once
  Arms: Cohort 1
Drug: Placebo — placebo to match 75 mg oral dose (prepared solution), given once
  Arms: Cohort 1
Drug: PF-04287881 — 150 mg oral dose (prepared solution) given once
  Arms: Cohort 2
Drug: Placebo — placebo to match 150 mg oral dose (prepared solution), given once
  Arms: Cohort 2
Drug: PF-04287881 — 300 mg oral dose (prepared solution) given once
  Arms: Cohort 3
Drug: Placebo — placebo to match 300 mg oral dose (prepared solution), given once
  Arms: Cohort 3
Drug: PF-04287881 — 750 mg oral dose (prepared solution) given once
  Arms: Cohort 4
Drug: Placebo — placebo to match 750 mg oral dose (prepared solution), given once
  Arms: Cohort 4
Drug: PF-04287881 — 1000 mg oral dose (prepared solution) given once
  Arms: Cohort 5
Drug: Placebo — placebo to match 1000 mg oral dose (prepared solution), given once
  Arms: Cohort 5
Drug: PF-04287881 — 1250 mg oral dose (prepared solution) given once
  Arms: Cohort 6
Drug: Placebo — placebo to match 1250 mg oral dose (prepared solution), given once
  Arms: Cohort 6
Drug: PF-04287881 — 1500 mg oral dose (prepared solution) given once
  Arms: Cohort 7
Drug: Placebo — placebo to match 1500 mg oral dose (prepared solution), given once
  Arms: Cohort 7
Drug: PF-04287881 — 300 mg oral dose (prepared solution) given once
  Arms: Cohort 8
Drug: Placebo — placebo to match 300 mg oral dose (prepared solution), given once
  Arms: Cohort 8
Drug: PF-04287881 — 750 mg oral dose (prepared solution) given once
  Arms: Cohort 9
Drug: Placebo — placebo to match 750 mg oral dose (prepared solution), given once
  Arms: Cohort 9
Drug: PF-04287881 — 1000 mg based on safety and PK from previous cohorts; oral dose (prepared solution) given once
  Arms: Cohort 10
Drug: Placebo — placebo to match 1000 mg oral dose (prepared solution), given once
  Arms: Cohort 10

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of PF-04287881 after a single oral dose in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers willing and able to be confined to the Clinical Research Unit and comply with study schedule.
* Women of non-childbearing potential only.
* Japanese subjects muct have 4 Japanese grandparents who were born in Japan.

Exclusion Criteria:

* Previous antibiotic use within 14 days prior to dosing.
* Use of antibiotics during hospitalization within 90 days prior to dosing.
* History of sensitivity to macrolides or ketolides.
* Presence of clinically significant eye conditions (other than corrective lenses).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of PF-04287881 after single oral dose. | Daily up to discharge, follow-up 7-10 days after dosing

SECONDARY OUTCOMES:
Pharmacokinetics of PF-04287881 after a single oral dose. | Pre-dose; Multiple timepoints on Day 1; 24, 36 hours Day 2; Single sample on Days 3-7.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0581001&StudyName=Safety%20And%20Pharmacokinetics%20Study%20Of%20PF-04287881%20In%20Healthy%20Adults